CLINICAL TRIAL: NCT00943033
Title: Toward Identifying the Mechanisms of Action in Mindfulness-Based Cognitive Therapy
Brief Title: Study of Mindfulness-Based Cognitive Therapy
Acronym: MBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Responsible Party: Principal Investigator, Sean Barnes, PhD, Binghamton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLI-FJVRF-08-SMB
Record Dates: First submitted 2009-07-13; First posted 2009-07-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Major Depressive Disorder
Keywords: MBCT; Mindfulness-Based Cognitive Therapy; Mindfulness; Meditation; Relapse Prevention; Recurrent Depression; Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy plus treatment as usual (Experimental)
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- MBCT Waitlist plus Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Mindfulness-Based Cognitive Therapy for the prevention of depressive relapse/recurrence
  Arms: Mindfulness-Based Cognitive Therapy plus treatment as usual

SUMMARY:
Research aimed at assessing changes in depressogenic thinking and the ability to disengage from depressogenic thinking following Mindfulness-Based Cognitive Therapy

ELIGIBILITY:
Inclusion Criteria:

* History of two or more Major Depressive Episodes or history of a Major Depressive Episode lasting at least one year
* Can speak, read, and understand English

Exclusion Criteria:

* Meet Criteria for Current Major Depressive Episode or are in partial remission
* BDI-II score above 19
* Abuse alcohol or drugs
* Current Dysthymic Disorder
* History of: psychosis when not depressed or intoxicated, Mania, Hypomania, Obsessive Compulsive Disorder, Posttraumatic Stress Disorder, Anorexia Nervosa, Bulimia Nervosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sustained Attention to Response Task | zero to four weeks pre-treatment and zero to three weeks post-treatment

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire | zero to four weeks pre-treatment and zero to three weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sean M. Barnes, MS, Principal Investigator — Binghamton University SUNY